CLINICAL TRIAL: NCT03504137
Title: A Pilot Study of Mobile Directly Observed Therapy (mDOT) for Immunosuppressant Adherence in Adolescent Kidney Transplant Recipients
Brief Title: A Pilot Study of mDOT for Immunosuppressant Adherence in Adolescent Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00168760
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-03

CONDITIONS: Medication Adherence; Kidney Transplant
Keywords: mHealth; kidney transplantation; medication adherence; video directly observed therapy
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: This is a single center prospective control trial. Participants in this study will use the mHealth application to manage and track their immunosuppression medical regimen post-transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Intervention (Experimental): Participants will receive the mHealth application either while they are an inpatient post-transplant, or at one of their post-transplant clinic visits. Study personnel will assist participants with downloading the mHealth application and explain its functioning. Participants will then use the application to aid in immunosuppressive medication adherence post-transplant.
  Interventions: Other: mHealth Intervention
- Standard of Care (No Intervention): Participants will not download the mHealth application. They will continue with their standard of care. Study personnel will send out surveys about general adherence. Participants will take their medications according to the instructions given by their transplant team and without any aid of the mHealth application.

INTERVENTIONS:
Other: mHealth Intervention — The video DOT app will allow transplant recipients to see their medication regimen, record themselves taking every dose, report side effects or symptoms, visualize their treatment progress, access educational content, and track appointments. This information is encrypted and transmitted to a HIPAA-secure web portal for providers to review.
  Arms: mHealth Intervention

SUMMARY:
The investigators are interested in whether or not the use of a mobile health (mHealth) application increases the rate of immunosuppression medication adherence among adolescent kidney transplant recipients. The investigators aim to test this by recruiting adolescent (ages 14-21) kidney transplant recipients to use an mHealth application to record themselves taking their immunosuppression medications, and tracking medication adherence over time. The study population will be approximately 50 adolescent kidney transplant recipients at the Johns Hopkins Hospital.

DETAILED DESCRIPTION:
In kidney transplant recipients, non-adherence to immunosuppressant medications post-transplant has been associated with a range of negative implications, including increased healthcare utilization, rejection of the graft, kidney loss, and death. Specifically, adolescents and young adults are the most at risk populations for experiencing death-censored graft loss and medication non-adherence. Previous studies have reported rates of non-adherence in this population ranging from 50-70%, and even minor deviations in immunosuppressant medication adherence have been shown to have negative effects. The use of mobile health (mHealth) technology could prove useful in aiding transplant recipients to stay adherent to their medical regimen.

We will use a mobile health platform that enables users to track dose-by-dose medication adherence through asynchronous, video directly observed therapy (DOT). This helps patients take their medication as prescribed and gives providers the assurance that their patients are supported and successful in treatment. DOT is the practice of watching a patient take every dose of medicine in-person, and has typically only been done in extreme cases because it can be both costly and burdensome: DOT is the standard of care for Tuberculosis treatment and has proven high-adherence rates. Through mHealth technology, DOT can be used more broadly and without added burden; emocha's technology allows this through enabling patients to use their mobile application to view their regimen, record themselves taking every dose of their medication, report side effects or symptoms, visualize their treatment progress, access educational content, and track appointments. This information is encrypted and transmitted to a HIPAA-secure web portal for providers to review. The aim of this study is to perform a pilot trial examining the rates of medication adherence in adolescent kidney transplant recipients who use a novel mHealth system, and to understand the acceptability/satisfaction with using this technology.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (14-21 years old)
* Have received a kidney transplant at the Johns Hopkins Hospital

Exclusion Criteria:

* Non-English speaking
* International

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
12-week immunosuppression medication adherence | 12 weeks
  After 12 weeks in the study, patients will complete the 4-item immunosuppressant therapy adherence instrument (ITAS) to determine self-reported medication adherence (scores range from 0-12 with 0 indicating very poor adherence and 12 indicating perfect adherence). Additionally, immunosuppression level trends will be tracked via electronic medical record review to determine medication adherence.

SECONDARY OUTCOMES:
Feasibility of using the mHealth Application as Assessed by a Semi-Structured Interview and a 17-Item Survey | 12 weeks
  After 12 weeks in the study, participants will be asked to participate in a semi-structured phone interview in which they will answer questions regarding their medication adherence habits and their thoughts on how our mHealth technology was or was not helpful. They will also complete a 17-question post-satisfaction survey assessing their satisfaction levels with the mhealth technology. Responses in the 17-item survey are on a 7-item Likert scale, ranging from Strongly Agree to Strongly Disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Macey L Henderson, JD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Geest S, Borgermans L, Gemoets H, Abraham I, Vlaminck H, Evers G, Vanrenterghem Y. Incidence, determinants, and consequences of subclinical noncompliance with immunosuppressive therapy in renal transplant recipients. Transplantation. 1995 Feb 15;59(3):340-7. PMID 7871562
- [Background] Butler JA, Roderick P, Mullee M, Mason JC, Peveler RC. Frequency and impact of nonadherence to immunosuppressants after renal transplantation: a systematic review. Transplantation. 2004 Mar 15;77(5):769-76. doi: 10.1097/01.tp.0000110408.83054.88. PMID 15021846
- [Background] Foster BJ, Dahhou M, Zhang X, Platt RW, Samuel SM, Hanley JA. Association between age and graft failure rates in young kidney transplant recipients. Transplantation. 2011 Dec 15;92(11):1237-43. doi: 10.1097/TP.0b013e31823411d7. PMID 22124283
- [Background] Douglas S, Blixen C, Bartucci MR. Relationship between pretransplant noncompliance and posttransplant outcomes in renal transplant recipients. J Transpl Coord. 1996 Jun;6(2):53-8. doi: 10.7182/prtr.1.6.2.x11r325882657x21. PMID 9188358
- [Background] Mehta P, Steinberg EA, Kelly SL, Buchanan C, Rawlinson AR. Medication adherence among adolescent solid-organ transplant recipients: A survey of healthcare providers. Pediatr Transplant. 2017 Nov;21(7). doi: 10.1111/petr.13018. Epub 2017 Jul 2. PMID 28670855
- [Background] Dobbels F, Van Damme-Lombaert R, Vanhaecke J, De Geest S. Growing pains: non-adherence with the immunosuppressive regimen in adolescent transplant recipients. Pediatr Transplant. 2005 Jun;9(3):381-90. doi: 10.1111/j.1399-3046.2005.00356.x. PMID 15910397
- [Background] Fredericks EM, Lopez MJ, Magee JC, Shieck V, Opipari-Arrigan L. Psychological functioning, nonadherence and health outcomes after pediatric liver transplantation. Am J Transplant. 2007 Aug;7(8):1974-83. doi: 10.1111/j.1600-6143.2007.01878.x. PMID 17617862
- [Background] Pai AL, McGrady M. Systematic review and meta-analysis of psychological interventions to promote treatment adherence in children, adolescents, and young adults with chronic illness. J Pediatr Psychol. 2014 Sep;39(8):918-31. doi: 10.1093/jpepsy/jsu038. Epub 2014 Jun 20. PMID 24952359
- [Background] Shaw RJ, Palmer L, Blasey C, Sarwal M. A typology of non-adherence in pediatric renal transplant recipients. Pediatr Transplant. 2003 Dec;7(6):489-93. doi: 10.1046/j.1397-3142.2003.00117.x. PMID 14870900
- [Background] De Geest S, Abraham I, Moons P, Vandeputte M, Van Cleemput J, Evers G, Daenen W, Vanhaecke J. Late acute rejection and subclinical noncompliance with cyclosporine therapy in heart transplant recipients. J Heart Lung Transplant. 1998 Sep;17(9):854-63. PMID 9773856
- [Background] Takemoto SK, Pinsky BW, Schnitzler MA, Lentine KL, Willoughby LM, Burroughs TE, Bunnapradist S. A retrospective analysis of immunosuppression compliance, dose reduction and discontinuation in kidney transplant recipients. Am J Transplant. 2007 Dec;7(12):2704-11. doi: 10.1111/j.1600-6143.2007.01966.x. Epub 2007 Sep 14. PMID 17868065
- [Background] Nahid P, Dorman SE, Alipanah N, Barry PM, Brozek JL, Cattamanchi A, Chaisson LH, Chaisson RE, Daley CL, Grzemska M, Higashi JM, Ho CS, Hopewell PC, Keshavjee SA, Lienhardt C, Menzies R, Merrifield C, Narita M, O'Brien R, Peloquin CA, Raftery A, Saukkonen J, Schaaf HS, Sotgiu G, Starke JR, Migliori GB, Vernon A. Official American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of America Clinical Practice Guidelines: Treatment of Drug-Susceptible Tuberculosis. Clin Infect Dis. 2016 Oct 1;63(7):e147-e195. doi: 10.1093/cid/ciw376. Epub 2016 Aug 10. PMID 27516382
- [Background] Chisholm MA, Lance CE, Williamson GM, Mulloy LL. Development and validation of the immunosuppressant therapy adherence instrument (ITAS). Patient Educ Couns. 2005 Oct;59(1):13-20. doi: 10.1016/j.pec.2004.09.003. PMID 16198214